CLINICAL TRIAL: NCT04877223
Title: Study of Blood Monocytes as a Predictive Marker of Cystic Fibrosis-related Bone Disease
Brief Title: Monocytes as Predictors of Cystic Fibrosis-related Bone Disease
Acronym: MucOs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-006-MucOs
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Bone disease; Monocytes; RANK; MCSF-R; Osteoclast
MeSH Terms: conditions — Cystic Fibrosis; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF: Patients with Cystic Fibrosis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Hypothesis: Circulating monocytes RANK and MCSF-R expression is predictive of Cystic Fibrosis-related Bone Disease.

Study design: Single-center comparative cross-sectional study Population: Patients with a CFTR channel mutation causing cystic fibrosis consulting the Centre de Ressources et de Compétences de la Mucoviscidose (CRCM) at Reims University Hospital will be recruited. Healthy controls will be recruited from donors at the Etablissement Français du Sang Grand Est, Reims.

Judgment criteria:

- Main judgment criterion: X Expression level of CD115 (MCSF receptor) and CD265 (RANK) evaluated by flow cytometry receptors on the membranes of circulating monocytes.

- Secondary judgment criteria: X Rate of circulating CD115 +, CD265 +, CD115 + / CD265 + monocytes X Number of multinucleated cells with more than 2 nuclei and with an actin ring observed under fluorescence microscopy after osteoclastic differentiation X Surface of dentin resorbed in vitro by osteoclasts during an osteoclastic functionality test on dentin X Serum S1P levels assayed by ELISA technique.

Investigation plan:

Any eligible patient will be offered to participate in the study during the consultation at the CRCM. If the patient agrees to participate in the study, he/she will be included. Participation in the study will not affect its coverage. Participation will lead to the collection of three tubes of whole blood additional to those used as part of usual care, as well as the collection of demographic data (age, sex, height, weight, body mass index), sports practice, clinical images and interpretation, medical history (diabetes, infectious status, bone metabolism disorders, drug treatments followed, psychiatric disorders). Any subsequent donor from the EFS GE collected under the ALC / PIL / DIR / AJR / FO / 606 agreement and presenting characteristics of age +/- 2 years and identical gender will then be included.

Statistical analysis plan:

Qualitative variables will be described in terms of number and percentage. The quantitative distribution variables according to the Normal law will be described in the form of mean +/- standard deviation or in the form of boxplots (median, quartiles, deciles) if a distribution not following the Normal law is observed. ANOVA test, non-parametric Wilcoxon signed-rank test or chi² test will be aplied depending on the application conditions. A value of p <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 and 65 years (+/- 2 years)
* Patients of the CRCM of Reims University Hospital
* Patients with at least one CF causing mutation in CFTR gene
* Patients agreeing to participate in the study (informed consent form)
* Patients fluent in French
* Patients affiliated with a social security regimen
* Healthy donors between 20 and 65 years (+/- 2 years)
* Healthy donors giving blood at EFS GE, Reims
* Healthy donors agreeing to participate in the study (informed consent form)
* Healthy donors fluent in French
* Healthy donors affiliated with a social security regimen
* Healthy donors whose characteristics agree with the ALC/PIL/DIR/AJR /FO/606 convention between EFS GE, Reims, and Reims Champagne-Ardenne University

Exclusion Criteria:

* Patient having a medical history that may compromise the protocol (psychiatric, medical or pharmacological disorders such as the use of anti-inflammatory drugs, or any compound that may alter or modify the inflammatory reaction in the week preceding the protocol).
* Pregnant or breastfeeding women
* Patient with eating disorders (anorexia, bulimia, overeating)
* Patient protected by law (guardianship, curatorship, hospitalized without their consent and not protected by law, deprived of liberty)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cystic fibrosis patients consulting the CRCM of Reims University Hospital. Healthy controls from Etablissement Français du Sang Grand Est, Reims
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of CD115 and CD265 expression on circulating monocytes | Immediately after sampling
  Flow cytometry

SECONDARY OUTCOMES:
Assessment of CD115+, CD265+ and CD115+/CD265+ cells | Immediately after sampling
  Flow cytometry
Count of multinucleated cells with actin ring | 3 weeks after sampling
  Phalloïdin/DAPI staining and microscope observation
Measurement of resorbed dentin surface | 3 weeks after sampling
  Scanning electron microscopy
Measurement of serum S1P concentration | Immediately after sampling
  ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Bruno RAVONINJATOVO, Principal Investigator — Centre de Ressources et de Compétences de la Mucoviscidose
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France